CLINICAL TRIAL: NCT00153829
Title: Chronic Illness Care Management (CICM) Study In Primary Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C. T. Lamont Primary Care Research Centre (Other)
Organization: Bruyère Health Research Institute. (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T-0528-029-22-CICM
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Illness; Quality of Life
Keywords: Chronic Disease; Quality of Life
MeSH Terms: conditions — Chronic Disease

INTERVENTIONS:
Behavioral: Multifaceted outreach facilitation for chronic illness care

SUMMARY:
The purpose of the study is to determine whether the quality of life of patients with multiple chronic conditions cared for by primary care physicians will improve due to the introduction of a chronic illness management intervention.

DETAILED DESCRIPTION:
There is international recognition for the need of introducing improvement in chronic illness care. However, primary care physicians face a host of challenges for providing the best possible care to their patients. One of these problems is the lack of proper administrative systems. There is evidence indicating that tailored out reach facilitation is an effective means to improve practice performance. Traditionally, the approach to care for chronically ill patients revolved mostly around the treatment of a specific chronic condition in an ad hoc basis. It is more common in family medicine for the patient to have several chronic conditions. There is also evidence showing that better health outcomes are obtained when the patients' life circumstances, desires and expectations are taken into consideration. Various models of chronic illness care have emerged that are patient center while attempting to be comprehensive. Our approach, following the Australian model, seeks to introduce systems/administrative innovations at the practice level, intended also to increase the involvement of patients with multiple chronic conditions on its own care, throw tailored out reach facilitation and care planning tools for physicians, in order to improve chronic illness management in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from any two or more chronic illnesses
* Patient should have been seen in the GP's office at least six to seven times in the previous year
* Patient should be 50 years of age or older

Exclusion Criteria:

* Suffering from dementia or a major psychiatric condition, being terminally ill, not being competent to give informed consent for participating in the study, or the doctors considers that the patient will not benefit from the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Difference between intervention and control groups of the average of the total SF-36 Health Survey physical and mental scores

SECONDARY OUTCOMES:
Difference between intervention and control groups of the average of the 'Healthy Days' Health Related Quality of Life-4 (HRQOL-4) scores

CONTACTS AND LOCATIONS:
Overall Officials: William Hogg, MD, CCFP, Principal Investigator — University of Ottawa; Jacques Lemelin, MD, CCFP, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Institute of Population Health, Ottawa, Ontario, Canada